CLINICAL TRIAL: NCT06934096
Title: Effects of Ultrasound Insonification of the Spleen on Platelet Activity and Coagulation Biomarkers in Healthy Human Subjects
Brief Title: Ultrasound of the Spleen Utilizing Low-energy (Diagnostic Level) Insonification.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-0307
Record Dates: First submitted 2025-04-02; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Hemostasis; Blood Biomarkers; Ultrasound
Keywords: Ultrasound of the spleen

STUDY DESIGN:
Intervention Model Description: Participants will be randomized from the three groups into two 30-minute stimulation sessions. One session will be active and the other sham. Participants are blinded to treatment group as well as the stimulation session.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focused insonification at enter of spleen (Experimental)
  Interventions: Device: Ultrasound Pulsed Doppler Imaging System
- Prolonged duration Insonification at center of spleen (Experimental)
  Interventions: Device: Ultrasound Pulsed Doppler Imaging System
- Prolonged insonification swept across the spleen (Experimental)
  Interventions: Device: Ultrasound Pulsed Doppler Imaging System

INTERVENTIONS:
Device: Ultrasound Pulsed Doppler Imaging System — Ultrasound pulsed doppler system accompanied with the abdominal curvilinear probe will be used for the purpose of collecting the data for the endpoints.

SUMMARY:
This is a three-cohort, randomized, double-blinded , sham-controlled, single-center, early feasibility research trial to determine whether organ-specific biologic effects on platelet activity and coagulation are achievable through selective ultrasound of the spleen utilizing low-energy (diagnostic-level) insonification.

* Group 1: Focused insonification at center of the spleen.
* Group 2: Prolonged duration insonification at center of the spleen
* Group 3: Prolonged duration insonification across the spleen.

Participants will receive 30 minutes of sham stimulation in the randomized group that is assigned to them, followed by active stimulation within the same group. Blood biomarkers (local and systemic) will be measured before and at several timepoints after stimulation to measure the molecular and cellular effects of the device

ELIGIBILITY:
Inclusion Criteria

1. Provision of signed and dated informed consent form
2. Willingness to comply with all study procedures and availability for the entire study duration
3. Male or female, aged 18 to 50 years
4. Individuals without physical disabilities or conditions/diseases that may make them incapable of undergoing the study procedure or otherwise places them at a greater risk of harm.
5. Individuals without significant past medical or surgical histories that would render them at a greater risk of harm
6. Individuals that are considered English Proficient due to the study requirements to follow verbal commands during the ultrasound session
7. Individuals that are considered active as assessed by type of activity (i.e., walking, running, etc.) and number of hours a week performing the various activities
8. Willing to adhere to the ultrasound study regimen
9. Individuals able to attend all study visits at approximately the same time of day (i.e., 8-12 pm)
10. Individuals able to comprehend the study goals and procedures, and can provide informed consent for participation

Exclusion Criteria:

1. Individuals participating in another research study that may affect the conduct or results of this study
2. Individuals considered substantially overweight or obese via body mass index (BMI > 30)
3. Individuals having or exhibiting any of the following:

   * surgery in the past 90 days
   * previous surgery of the spleen or splenectomy, esophagus, lungs, stomach, duodenum, or liver
   * recent traumatic injury, including intracerebral hemorrhage and visceral injury
   * end stage renal disease and/or uremia
   * active malignancy
   * previous leukemia and/or lymphoma
   * human immunodeficiency virus infection or AIDS
   * rheumatoid arthritis or other immune-mediated diseases (e.g. inflammatory bowel disease)
   * arrhythmias, including but not limited to, atrial fibrillation, atrial flutter, clinically significant bradycardia, ventricular arrhythmias, and A-V block
   * implanted pacemaker or cardioverter/defibrillator (AICD)
   * history of stable or unstable angina, myocardial infarction, angioplasty, or coronary arterial by-pass grafting surgery
   * history of stroke or TIA
   * history of deep venous thrombosis (DVT) and/or pulmonary embolism (PE)
   * previous episodes of pancreatitis
   * spinal disorders
   * chronic pain syndromes
   * stage III-IV pressure ulcers
   * sickle cell anemia or other anemia syndromes
   * diagnosed with fever of unknown origin (FUO)
   * previously or currently implanted vagus nerve stimulator
   * previously or currently implanted spinal cord stimulator or other chronically implanted electronic medical device
   * history of seizures
   * history of cancer
4. Individuals who have taken any of the following medications within two weeks of receiving ultrasound delivery:

   * anti-coagulants (warfarin, Xarelto)
   * anti-platelet agent (aspirin, clopidogrel)
   * anti-inflammatory (aspirin, NSAIDs)
   * anti-hypertensive (α-methyldopa)
   * epinephrine-related drugs, norepinephrine-related drugs, and drugs that stimulate release of epinephrine and/or norepinephrine (Micronefrin, Asthmanefrin)
   * immunosuppressive agents (steroids, newer immunomodulatory drugs)
   * alpha and/or beta-adrenoceptor blocking agents
   * anti-seizure medications
   * other medications, supplements, etc. that may interfere with the ultrasound delivery or study results
5. Individuals with a substance abuse (alcoholism or other) problem
6. Individuals that consumed alcohol within 7 days of the baseline visit
7. Individuals currently using or have used cocaine, heroin, marijuana, or other illicit recreational drugs within the past 3 months
8. Prisoners
9. Participant has a history of thrombocytopenia (platelet count <100k)
10. Participant has reported coagulopathy (elevated PT, PTT, elevated activated clotting time (ACT))
11. Participant has internal bleeding, external bleeding, easy bruising
12. Participant has a history of abnormal bleeding or blood disorder, including anemia or anemia-related disorders
13. Participant has a history of thrombocytopenia (platelet count <100k)
14. Participant has a history of coagulopathy, including hemophilia, stroke, pulmonary embolism, myocardial infarction, or deep vein thromboses
15. Participant has a history of conditions that can cause coagulopathic conditions, including atrial fibrillation, heart valve surgery or replacement, hip or knee replacement, or clotting disorders
16. Participants using coagulation- or platelet-modifying therapies such as clotting factor products, emicizumab, desmopressin acetate, epsilon amino caproic acid, heparin and its derivatives, argatroban, desirudin, bivalirudin, dabigatran, apixaban, edoxaban, betrixaban
17. Participant has a history of chronic tobacco use or has ingested nicotine via smoking, vaping, smokeless tobacco, or nicotine patches in the past three months
18. Participant has consumed caffeine within the past 12 hours
19. Participant has received a blood transfusion within 30 days prior to study
20. Participant has a history of neurologic diseases or traumatic brain injury
21. Women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study
22. Females who are pregnant, lactating or menstruating
23. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants are risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-21 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether diagnostic-level ultrasound to the spleen can modulate systemic blood biomarkers of hemostasis | 4 hours
  The primary objective is to determine whether diagnostic-level ultrasound to the spleen can modulate systemic blood biomarkers of hemostasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States